CLINICAL TRIAL: NCT06904222
Title: A Phase I, Randomized, Observer-blinded, Placebo-Controlled, Dose Escalation Clinical Trial to Assess the Safety and Immunogenicity of the Respiratory Syncytial Virus (RSV) Vaccine, LYB005 in Adults Aged 18 Years and Older
Brief Title: Safety and Immunogenicity of the Recombinant Respiratory Syncytial Virus (RSV) Vaccine in Adults Aged 18 Years and Older
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LYB005/CT-CHN-101
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: Respiratory Syncytial Virus; Acute Respiratory Infection; Lower Respiratory Track Disease
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in one of six cohorts, including Cohort 1 (18-59 years, low dose, n=15), Cohort 2 (18-59 years, middle dose, n=15), Cohort 3 (≥60 years, low dose, n=15), Cohort 4 (18-59 years, high dose, n=15), Cohort 5 (≥60 years, middle dose, n=15), and Cohort 6 (≥60 years, high dose, n=15). In each cohort, five sentinels were set up, and they were randomly vaccinated with the investigational vaccine without A01B adjuvant, the investigational vaccine with A01B adjuvant, or placebo in a 2:2:1 ratio. The remaining participants were randomly vaccinated in a 2:2:1 ratio with the investigational vaccine without A01B adjuvant, the investigational vaccine with A01B adjuvant, or placebo. For both sentinels and remaining participants, the investigational vaccine group and the control group (placebo) are enrolled parallelly.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Low dose antigen of LYB005 without A01B adjuvant (Experimental): Subjects aged 18 years and older will be vaccinated with 1 dose of LYB005 (low dose antigen without A01B adjuvant) at Day 0.
  Interventions: Biological: Low dose antigen of LYB005 without A01B adjuvant
- Low dose antigen of LYB005 with A01B adjuvant (Experimental): Subjects aged 18 years and older will be vaccinated with 1 dose of LYB005 (low dose antigen with A01B adjuvant) at Day 0.
  Interventions: Biological: Low dose antigen of LYB005 with A01B adjuvant
- Middle dose antigen of LYB005 without A01B adjuvant (Experimental): Subjects aged 18 years and older will be vaccinated with 1 dose of LYB005 (middle dose antigen without A01B adjuvant) at Day 0.
  Interventions: Biological: Middle dose antigen of LYB005 without A01B adjuvant
- Middle dose antigen of LYB005 with A01B adjuvant (Experimental): Subjects aged 18 years and older will be vaccinated with 1 dose of LYB005 (middle dose antigen with A01B adjuvant) at Day 0.
  Interventions: Biological: Middle dose antigen of LYB005 with A01B adjuvant
- High dose antigen of LYB005 without A01B adjuvant (Experimental): Subjects aged 18 years and older will be vaccinated with 1 dose of LYB005 (high dose antigen without A01B adjuvant) at Day 0.
  Interventions: Biological: High dose antigen of LYB005 without A01B adjuvant
- High dose antigen of LYB005 with A01B adjuvant (Experimental): Subjects aged 18 years and older will be vaccinated with 1 dose of LYB005 (high dose antigen with A01B adjuvant) at Day 0.
  Interventions: Biological: High dose antigen of LYB005 with A01B adjuvant
- Placebo (Placebo Comparator): Subjects aged 18 years and older will be vaccinated with 1 dose of placebo at Day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose antigen of LYB005 without A01B adjuvant — 0.5 mL per dose, containing a total of 30 μg antigen without A01B adjuvant.
  Arms: Low dose antigen of LYB005 without A01B adjuvant
Biological: Low dose antigen of LYB005 with A01B adjuvant — 0.5 mL per dose, containing a total of 30 μg antigen adjuvanted with A01B.
  Arms: Low dose antigen of LYB005 with A01B adjuvant
Biological: Middle dose antigen of LYB005 without A01B adjuvant — 0.5 mL per dose, containing a total of 60 μg antigen without A01B adjuvant.
  Arms: Middle dose antigen of LYB005 without A01B adjuvant
Biological: Middle dose antigen of LYB005 with A01B adjuvant — 0.5 mL per dose, containing a total of 60 μg antigen adjuvanted with A01B.
  Arms: Middle dose antigen of LYB005 with A01B adjuvant
Biological: High dose antigen of LYB005 without A01B adjuvant — 0.5 mL per dose, containing a total of 120 μg antigen without A01B adjuvant.
  Arms: High dose antigen of LYB005 without A01B adjuvant
Biological: High dose antigen of LYB005 with A01B adjuvant — 0.5 mL per dose, containing a total of 120 μg antigen adjuvanted with A01B.
  Arms: High dose antigen of LYB005 with A01B adjuvant
Biological: Placebo — 0.5 mL 0.9% sodium chloride (normal saline) injection per dose
  Arms: Placebo

SUMMARY:
This phase 1 study in China will evaluate the safety and immunogenicity of the the Respiratory Syncytial Virus (RSV) Vaccine, LYB005 in adults aged 18 years and older.

DETAILED DESCRIPTION:
A randomized, observer-blinded, placebo-controlled, dose escalation trial will be conducted to observe the safety and immunogenicity of LYB005 in adults aged 18 years and older. A total of 90 healthy subjects will be enrolled and stratified by age (18-59 years and ≥60 years in a 1:1 ratio). Six formulations of LYB005 will be provided, three dose levels of antigen with or without A01B adjuvant.

A sentinel and escalating dosing approach will be used for close monitoring of safety to minimize risk to participants. Participants will be enrolled in one of six cohorts, including Cohort 1 (18-59 years, low dose, n=15), Cohort 2 (18-59 years, middle dose, n=15), Cohort 3 (≥60 years, low dose, n=15), Cohort 4 (18-59 years, high dose, n=15), Cohort 5 (≥60 years, middle dose, n=15), and Cohort 6 (≥60 years, high dose, n=15). In each cohort, five sentinels were set up, and they were randomly vaccinated with the investigational vaccine without A01B adjuvant, the investigational vaccine with A01B adjuvant, or placebo in a 2:2:1 ratio. The remaining participants were randomly vaccinated in a 2:2:1 ratio with the investigational vaccine without A01B adjuvant, the investigational vaccine with A01B adjuvant, or placebo. A single-dose immunization schedule will be adopted.

ELIGIBILITY:
Inclusion Criteria:

1. Residents aged 18 years and older (at the time of screening), regardless of gender;
2. Participants can provide valid identification, voluntarily agree to participate in the study, and sign the Informed Consent Form, and are able to attend all planned follow-up visits and comply with the protocol requirements;
3. Axillary temperature < 37.3°C on the day of enrollment;
4. Females of childbearing potential should use effective contraceptive measures one month before enrollment; females of childbearing potential (excluding those who have undergone tubal ligation, bilateral oophorectomy, or hysterectomy) and male participants should practice effective contraception and avoid pregnancy plans, as well as sperm or egg donation plans from the time of enrollment until 6 months after the full course of vaccination. Effective contraceptive methods include oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release local contraceptives, contraceptive patches, intrauterine devices, sterilization, abstinence, condoms, diaphragms, cervical caps, etc.

Exclusion Criteria:

1. Allergy to the investigational vaccine or its excipients, or a history of anaphylactic shock or other serious adverse reactions to other vaccines;
2. Previous vaccination against Respiratory Syncytial Virus;
3. A confirmed diagnosis or etiological evidence of respiratory syncytial virus infection and related diseases caused by the infection within 12 months before enrollment;
4. Has taken antipyretics, analgesics or anti-allergy drugs within 24 hours before enrollment;
5. Has received any vaccine within 14 days before vaccination, or have received a live vaccine within 28 days;
6. Has received blood or blood-related products, including immunoglobulin, within 3 months prior to enrollment; or plan to use them during the study period;
7. Individual with the following diseases:

   * Has acute diseases or are in the acute exacerbation period of chronic diseases within 3 days before vaccination;
   * Diagnosed with congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
   * History of congenital or acquired immunodeficiency or autoimmune diseases;
   * Chronic administration (≥14 consecutive days) of corticosteroids (dose ≥ 20 mg/day prednisone or equivalent dose) or other immunosuppressants within the past 3 months, with the exception of inhaled or topical steroids, or short-term use (<14 consecutive days) of oral corticosteroids;
   * Neurological diseases or family history (seizures, epilepsy, encephalopathy, etc.); history of psychiatric disorders or family history;
   * Asplenia or functional asplenia;
   * Severe or uncontrolled or hospitalization-required cardiovascular diseases, diabetes, blood and lymphatic system diseases, immune system diseases, liver and kidney diseases, respiratory system diseases, metabolic and skeletal system diseases, or malignant tumors;
   * Contraindications for intramuscular injection and blood drawing, such as coagulation disorders, thrombosis or hemorrhagic diseases, or situations requiring continuous use of anticoagulants;
   * Severe hypertension that cannot be controlled by medication (measured on-site: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
8. History of major surgery within 12 weeks prior to enrollment (as determined by the investigator), or not fully recovered from the surgery, or having plans for major surgery during the anticipated period of the subject's participation in the study;
9. History of long-term alcohol abuse and/or drug abuse;
10. Individual who is currently participating in other research or unregistered product (drugs, vaccines, or devices, etc.) clinical studies, or plan to participate in other clinical studies before the end of this clinical study;
11. Other conditions that may impact the subject's safety or influence the assessment of vaccine response, as determined by the investigator;
12. Exclusion criteria for specific populations: lactating or pregnant women during the clinical research period, or women of childbearing age with a positive pregnancy test before vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of immediate adverse events | Within 30 minutes after vaccination
  The incidence and severity of any adverse events (AEs) within 30 minutes after vaccination
Incidence of solicited AE | Within 0-7 days after vaccination
  Occurrence and severity of solicited local injection site reactions for 7 days (Day 0-Day 7) following vaccination. (i.e., pain, redness, swelling).
  Occurrence and severity of solicited systemic reactions for 7 days (Day 0-Day 7) following vaccination. (i.e., myalgia, fatigue, headache, chills, fever).
Incidence of unsolicited AEs | Within 28 days after vaccination
  The incidence and severity of any unsolicited AEs, including all AEs, except solicited AEs reported Days 0~28 after the vaccination.
Incidence of clinically significant abnormalities in clinical laboratory tests | 3 days after vaccination
  The incidence of clinically significant abnormalities in clinical laboratory tests (hematology, blood chemistry, coagulation function, and urinalysis) on Day 3 after vaccination.
Occurrence of serious adverse events (SAEs) and adverse events of special interests (AESIs) | 12 months after vaccination
  The incidence of any SAEs and AESIs from the first vaccination up to 12 months after vaccination.

SECONDARY OUTCOMES:
The geometric mean titer (GMT) of Neutralizing Antibodies Against RSV A and RSV B | 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Measured by microneutralization assay.
Geometric Mean Fold Rise (GMFR) for Neutralizing Antibodies Against RSV A and RSV B | 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Change from prevaccination in geometric mean fold rise of Neutralizing antibody titer Against RSV A and RSV B
The geometric mean concentration (GMC) for Pre-fusion Protein Specific Binding Antibodies | 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA).
Number of Pre-fusion Protein Specific Interferon-gamma and Interleukin-4 spot-forming cells | 28 days after vaccination
  T-cell responses to vaccine antigen in peripheral blood mononuclear cells (PBMCs) determined by enzyme-linked immunosorbent spot (ELISpot).

CONTACTS AND LOCATIONS:
Overall Officials: Beifang Yang, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Dangyang City Center for Disease Control and Prevention, Dangyang, China

IPD SHARING:
Plan to Share IPD: No